CLINICAL TRIAL: NCT05665569
Title: Effects of Flourish HEC Vaginal Care System in Postpartum Women Undergoing Pelvic Physical Therapy for Birth-Related Pelvic Floor Disorders
Brief Title: Effects of Flourish HEC Vaginal Care System on Birth-Related Pelvic Floor Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vaginal Biome Science (Other)
Collaborators: Empower Yourself PT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPT0922
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Floor Disorders
Keywords: vaginal microbiome; vaginal pH
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine Care (Active Comparator): Women will undergo routine pelvic physical therapy for birth-related pelvic floor disorders as determined by their physical therapist who is also the Principal Investigator.
  Interventions: Other: Routine pelvic physical therapy
- Flourish HEC (Experimental): In addition to routine physical therapy, women will use a 3-component vaginal hygiene system, "Flourish HEC" (HEC = hydroxyethylcellulose to differentiate this system from a prior Flourish system based in aloe) plus a personal lubricant called BioNude.
  Interventions: Device: Flourish HEC, which contains BioNourish; Other: Routine pelvic physical therapy

INTERVENTIONS:
Device: Flourish HEC, which contains BioNourish — The Flourish HEC vaginal hygiene system comprises Balance intimate wash used daily, BioNourish vaginal moisturizing gel used daily, and BiopHresh homeopathic vaginal suppository containing probiotics, used once every 3 days. In addition, for all therapy requiring insertion in the clinic or at home, or for sex if desired, BioNude personal lubricant will be used. These four products are intended to allow the vaginal microbiome to self-correct by supporting the vaginal environment in terms of providing pH, osmolality, and lactic acid levels that match those in a healthy vagina.
  Arms: Flourish HEC
Other: Routine pelvic physical therapy — Routine pelvic physical therapy may include external and internal manual techniques, exercises, diaphragmatic breathing exercises, and other modalities.

SUMMARY:
The goal of this clinical trial is to learn about how the vaginal microbiome affects pelvic floor disorders in women who have recently given birth. The main question it aims to answer is:

• Can improving the vaginal microbiome allow women to improve muscle strength, improve muscle tone, and reduce tissue inflammation faster than women who do not use a vaginal hygiene system to improve their microbiome?

Over a 3-month period, participants will be assessed three times for:

* vaginal microbiome
* vaginal pH
* pelvic muscle strength
* pelvic muscle tension
* vulvovaginal tissue color At each of these 3 assessments, women will answer questions on a questionnaire. Half of the women will be asked to use a vaginal hygiene system at home during these 3 months.

Researchers will compare use of a three-product vaginal hygiene system plus a specific vaginal lubricant to see if using these products improves the vaginal microbiome and the pelvic floor outcomes listed above.

DETAILED DESCRIPTION:
The vaginal microbiome interacts with vaginal epithelial cells and host immune cells in varying ways depending on the presence of particular species. Presence of high quantities of Lactobacillus species, which are considered healthy, downregulate pro-inflammatory markers and upregulate anti-inflammatory markers. On the other hand, BV-associated bacteria such as Gardnerella vaginalis, Atopobium (Fannyhessea) vaginae, Prevotella bivia, Mobiluncus curtisii and others are associated with increased pro-inflammatory markers and reduced anti-inflammatory molecules. The investigators predict that improving the vaginal microbiome by using an over-the-counter vaginal care system will increase levels of Lactobacillus species, reduce levels of BV-associated bacteria, and reduce overall tissue inflammation, thereby speeding tissue healing.

The original Flourish® Vaginal Care System, with slightly different vaginal moisturizer (with aloe), has recently been shown in a clinical study to reduce vaginal pH from 4.81 (unhealthy, elevated) to 4.05 (healthy) and prevent recurrence of bacterial vaginosis over a 10-week study period. The proposed study uses a newly formulated product that is gentler (no aloe) because the study population is likely to have high sensitivity based on inclusion criteria involving tissue trauma.

Pelvic floor disorders (or pelvic floor dysfunction) affect a large percentage of females around the globe that may manifest as vulvovaginal pain, pelvic/bladder pain, urinary or fecal incontinence, pelvic organ prolapse, urinary urgency, urinary frequency, and much more. It can take on several forms, including either weakness of pelvic floor muscles (causing incontinence or prolapse), or excessive tightness (hypertonia) of the same muscles; sometimes these occur simultaneously in the same individual. Pelvic floor disorders can significantly disrupt daily life, for example causing patients to wake up multiple times in the night to urinate, or causing leakage of urine or feces at inopportune times, causing women to make dramatic changes to their lives to avoid embarrassing situations or pain. In addition, incontinence may be responsible for urinary tract and vaginal infections.

Women who have given birth vaginally often experience trauma to the pelvic floor that results in pelvic floor disorders. They often seek treatment from physical therapists, which may begin as early as six weeks after delivery or may not occur until years after the initial trauma. Pelvic physical therapy interventions can include exercises, diaphragmatic breathing techniques, external and internal manual techniques, and other modalities to improve muscle strength, muscle tension, tissue inflammation, and reduce degree of symptoms.

Pelvic physical therapy often involves manual techniques such as myofascial release, soft tissue mobilization, and scar tissue mobilization in conjunction with dilator use at home to reduce tension in the muscles of the pelvic floor muscles. Lubricants are typically used on the finger or device to ease insertion. However, many lubricants, including some of those used clinically, have been shown to cause excessive exfoliation of vaginal epithelial cells and to induce dysbiosis. The most damaging lubricants are those that are hyperosmolar and those which contain specific antimicrobial ingredients, such as nonoxynol-9, chlorhexidine gluconate, polyquaternium-15, and parabens. The investigators hypothesize that use of lubricants such as these increase inflammation in the vagina, slowing the rate of progress in physical therapy and possibly causing conditions such as bacterial vaginosis, aerobic vaginitis, or vaginal yeast infections. The investigators predict that using a lubricant designed to closely match healthy vaginal secretions, along with a hygiene system that promotes healthy flora, will enable pelvic physical therapy patients to improve more quickly and/or more completely without complications. The investigators also hypothesize that there may be specific microbiome patterns observed in women with this type of pelvic floor disorder that are distinct from healthy women.

Together, it is hypothesized that using a specific over-the-counter commercially available vaginal hygiene system plus lubricant which have all been formulated with vaginal tissue and microbiome health in mind will improve the vaginal microbiome and help postpartum women achieve their pelvic physical therapy goals faster and/or more thoroughly.

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18
2. Vaginal delivery within the past year
3. Attending a pelvic physical therapy clinic treatment of birth-related pelvic floor disorder with one or more of the following symptoms: vulvovaginal pain, pelvic/bladder pain, urinary or fecal incontinence, or dyspareunia.
4. Needing approximately three months of treatment sessions

Exclusion Criteria:

1. Known allergies or sensitivities to any ingredients of the Flourish HEC Vaginal Care System
2. Immunosuppressed or otherwise immunocompromised
3. Vaginal infection at the start of the study other than bacterial vaginosis or yeast infection (these may be treated prior to starting the protocol)
4. Current use of any antibiotics
5. Surgery within the past 3 months
6. Pregnant or trying to conceive during the trial
7. Recent (within past 6 months) usage of any Good Clean Love products
8. Psychiatric/mental disorders triggered by questions related to vulvar or vaginal health, by pelvic exams

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Changes in vaginal microbiome over time | Baseline to 6 weeks
  Vaginal microbiome composition will be assessed by whole-genome sequencing at three timepoints; this outcome assesses the initial 6-week time period. Individual biomes will be categorized as healthy, intermediate, or unhealthy using the VALENCIA model to assign community state types (CSTs). CSTs I, II, and V are "healthy"; CST III is "intermediate"; CST IV is "unhealthy". Changes over time will be analyzed by Krusal-Wallis.
Changes in vaginal microbiome over time | Baseline to 3 months
  Vaginal microbiome composition will be assessed by whole-genome sequencing at three timepoints; this outcome assesses the entire duration of the study. Individual biomes will be categorized as healthy, intermediate, or unhealthy using the VALENCIA model to assign community state types (CSTs). CSTs I, II, and V are "healthy"; CST III is "intermediate"; CST IV is "unhealthy". Changes over time will be analyzed by Krusal-Wallis.
Changes in vaginal pH over time | Baseline to 6 weeks
  Vaginal pH will be assessed using colorimetric pH test strips at three timepoints; this outcome assesses the initial 6-week period. Data will be analyzed by repeated measures ANOVA.
Changes in vaginal pH over time | Baseline to 3 months
  Vaginal pH will be assessed using colorimetric pH test strips at three timepoints; this outcome assesses the entire study duration. Data will be analyzed by repeated measures ANOVA.

SECONDARY OUTCOMES:
Changes in pelvic floor muscle strength over time | Baseline to 6 weeks
  Changes in pelvic floor muscle strength will be assessed by vaginal palpation using the Modified Oxford Grading System, a Likert scoring system on a scale of 0 to 5, with 0 being no contraction, and 5 being strong contraction. This outcome assesses the initial 6-week period. Data will be analyzed by Kruskal-Wallis.
Changes in pelvic floor muscle strength over time | Baseline to 3 months
  Changes in pelvic floor muscle strength will be assessed by vaginal palpation using the Modified Oxford Grading System, a Likert scoring system on a scale of 0 to 5, with 0 being no contraction, and 5 being strong contraction. This outcome assesses the entire study duration. Data will be analyzed by Kruskal-Wallis.
Changes in pelvic floor muscle tension over time | Baseline to 6 weeks
  Changes in pelvic floor muscle tension will be assessed by vaginal palpation using a Likert scoring system on a scale of 0 to 5, with 0 being no muscle tension, and 5 being high muscle tension. This outcome assesses the initial 6-week period. Data will be analyzed by Kruskal-Wallis.
Changes in pelvic floor muscle tension over time | Baseline to 3 months
  Changes in pelvic floor muscle tension will be assessed by vaginal palpation using a Likert scoring system on a scale of 0 to 5, with 0 being no muscle tension, and 5 being high muscle tension. This outcome assesses the entire study duration. Data will be analyzed by Kruskal-Wallis.
Changes in vulvovaginal tissue inflammation over time | Baseline to 6 weeks
  Changes in vulvovaginal tissue inflammation will be assessed by assigning tissue color using a Likert scoring system on a scale of 0 to 3, with 0 being blanched tissue, 1 being healthy pink tissue, 2 being dark pink, and 3 being red inflamed tissue. This outcome assesses the initial 6-week period. Data will be analyzed by Kruskal-Wallis.
Changes in vulvovaginal tissue inflammation over time | Baseline to 3 months
  Changes in vulvovaginal tissue inflammation will be assessed by assigning tissue color using a Likert scoring system on a scale of 0 to 3, with 0 being blanched tissue, 1 being healthy pink tissue, 2 being dark pink, and 3 being red inflamed tissue. This outcome assesses the entire study duration. Data will be analyzed by Kruskal-Wallis.
Changes in vulvovaginal symptoms over time | Baseline to 6 weeks
  Changes in vulvovaginal symptoms will be assessed by questionnaires using either yes/no (Vulvovaginal Symptoms Questionnaire) or Likert-based scoring (scale of 0 to 3, where 0 is no symptom and 3 is severe or all the time). This outcome assesses the initial 6-week period. Data will be analyzed by Mann-Whitney U or Kruskal-Wallis as appropriate per question.
Changes in vulvovaginal symptoms over time | Baseline to 3 months
  Changes in vulvovaginal symptoms will be assessed by questionnaires using either yes/no (Vulvovaginal Symptoms Questionnaire) or Likert-based scoring (0 to 3, with 0 being no symptom and 3 being severe or all the time). This outcome assesses the entire study duration. Data will be analyzed by Mann-Whitney U or Kruskal-Wallis as appropriate per question.
Time to resolution of most bothersome symptom (MBS) | Baseline to 3 months
  Each participant's MBS will be tracked to determine which week of the study the participant no longer reported experiencing that symptom. Time to resolution of the MBS will be analyzed by Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kowenski, DPT, Principal Investigator — Empower Yourself PT
Locations (1):
- Empower Yourself PT, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chidawanyika T, Yi CHC, Kelly-Martin R, Cleland J, DuPriest E. Clinical trial to survey results of Flourish vaginal care system for recurrent BV [A80]. Obstet Gynecol. 2022;139:24S. doi:10.1097/01.AOG.0000826648.49549.01
- [Background] World Health Organization. Use and Procurement of Additional Lubricants for Male and Female Condoms: WHO/UNFPA/FHI360 Advisory Note.; 2012:1-8.
- [Background] Laniewski P, Herbst-Kralovetz MM. Bacterial vaginosis and health-associated bacteria modulate the immunometabolic landscape in 3D model of human cervix. NPJ Biofilms Microbiomes. 2021 Dec 13;7(1):88. doi: 10.1038/s41522-021-00259-8. PMID 34903740
- [Background] France MT, Ma B, Gajer P, Brown S, Humphrys MS, Holm JB, Waetjen LE, Brotman RM, Ravel J. VALENCIA: a nearest centroid classification method for vaginal microbial communities based on composition. Microbiome. 2020 Nov 23;8(1):166. doi: 10.1186/s40168-020-00934-6. PMID 33228810
- [Background] Dezzutti CS, Brown ER, Moncla B, Russo J, Cost M, Wang L, Uranker K, Kunjara Na Ayudhya RP, Pryke K, Pickett J, Leblanc MA, Rohan LC. Is wetter better? An evaluation of over-the-counter personal lubricants for safety and anti-HIV-1 activity. PLoS One. 2012;7(11):e48328. doi: 10.1371/journal.pone.0048328. Epub 2012 Nov 7. PMID 23144863
- [Background] Wilkinson EM, Laniewski P, Herbst-Kralovetz MM, Brotman RM. Personal and Clinical Vaginal Lubricants: Impact on Local Vaginal Microenvironment and Implications for Epithelial Cell Host Response and Barrier Function. J Infect Dis. 2019 Nov 6;220(12):2009-2018. doi: 10.1093/infdis/jiz412. PMID 31539059
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Ananthapadmanabhan KP, Moore DJ, Subramanyan K, Misra M, Meyer F. Cleansing without compromise: the impact of cleansers on the skin barrier and the technology of mild cleansing. Dermatol Ther. 2004;17 Suppl 1:16-25. doi: 10.1111/j.1396-0296.2004.04s1002.x. PMID 14728695